CLINICAL TRIAL: NCT07394582
Title: Preoperative Optimization Before Total Hip or Knee Replacement Surgery - a Controlled, Randomized, Single-blind Study
Brief Title: Preoperative Optimization Before Total Hip or Knee Replacement Surgery
Acronym: PrOpE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EK-Nr. 1193/2025
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Prehabilitation; Preoperative Care
Keywords: Preoperative Optimization; orthopedic surgery
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, single blinded (patient-blinded) with two study groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Group (No Intervention): Participants receive usual medical care before and after surgery.
- Intervention Group (Experimental): In addition to standard care, participants receive an individualised preparation programme over several weeks before surgery. This programme may include:
  * Personalised physical exercise
  * Nutritional assessment and advice
  * Support for stress, pain, and mental well-being
  * Review of regular medications
  Interventions: Other: Prehabilitation

INTERVENTIONS:
Other: Prehabilitation — * Personalised physical exercise
  * Nutritional assessment and advice
  * Support for stress, pain, and mental well-being
  * Review of regular medications Some elements may be delivered at home or via telemedicine, depending on individual needs.
  Arms: Intervention Group

SUMMARY:
Preoperative Optimisation prior to Hip and Knee Arthroplasty (PrOpE) Many patients scheduled for planned hip or knee replacement surgery have health conditions that may affect recovery, such as reduced physical fitness, nutritional problems, multiple medications, or increased stress and anxiety. These factors can increase the risk of complications and delay recovery after surgery.

The PrOpE study examines whether a structured preparation programme before surgery, known as preoperative optimization or prehabilitation, can be safely implemented and may support recovery after hip or knee replacement.

Aim of the study The main aim is to assess the feasibility of a comprehensive preoperative optimisation programme and to explore its potential effects on recovery and health outcomes. The results will help improve future care for patients undergoing major orthopaedic surgery.

Who can participate? Adult patients scheduled for elective total hip or knee replacement surgery who are classified as ASA >2, aged between 18 and 99 years old and without a severe cognitive impairment. Participation is voluntary.

Study design

A total of 180 participants will be included and randomly assigned to one of two groups:

• Standard Care Group: Participants receive usual medical care before and after surgery.

• Intervention Group:

In addition to standard care, participants receive an individualised preparation programme over several weeks before surgery. This programme may include:

* Personalised physical exercise
* Nutritional assessment and advice
* Support for stress, pain, and mental well-being
* Review of regular medications Some elements may be delivered at home or via telemedicine, depending on individual needs.

What information is collected? The study evaluates recovery after surgery, including complications, length of hospital stay, physical function, quality of life, and use of health care services. Questionnaires, physical tests, and blood samples are used to better understand health status before and after surgery.

Risks and benefits The study involves low additional risk. All measures are adapted to individual abilities and supervised by trained professionals. The main burden is the additional time required for participation. Participants in the optimisation group may benefit from improved preparation for surgery. The study also contributes to improving care for future patients.

DETAILED DESCRIPTION:
Preoperative Optimisation prior to Hip and Knee Arthroplasty (PrOpE) Many patients scheduled for planned hip or knee replacement surgery have health conditions that may affect recovery, such as reduced physical fitness, nutritional problems, multiple medications, or increased stress and anxiety. These factors can increase the risk of complications and delay recovery after surgery.

The PrOpE study examines whether a structured preparation programme before surgery, known as preoperative optimization or prehabilitation, can be safely implemented and may support recovery after hip or knee replacement.

Aim of the study The main aim is to assess the feasibility of a comprehensive preoperative optimisation programme and to explore its potential effects on recovery and health outcomes. The results will help improve future care for patients undergoing major orthopaedic surgery.

Who can participate? Adult patients scheduled for elective total hip or knee replacement surgery who are classified as ASA >2, aged between 18 and 99 years old and without a severe cognitive impairment. Participation is voluntary.

Study design

A total of 180 participants will be included and randomly assigned to one of two groups:

• Standard Care Group: Participants receive usual medical care before and after surgery.

• Intervention Group:

In addition to standard care, participants receive an individualised preparation programme over several weeks before surgery. This programme may include:

* Personalised physical exercise
* Nutritional assessment and advice
* Support for stress, pain, and mental well-being
* Review of regular medications Some elements may be delivered at home or via telemedicine, depending on individual needs.

What information is collected? The study evaluates recovery after surgery, including complications, length of hospital stay, physical function, quality of life, and use of health care services. Questionnaires, physical tests, and blood samples are used to better understand health status before and after surgery.

Risks and benefits The study involves low additional risk. All measures are adapted to individual abilities and supervised by trained professionals. The main burden is the additional time required for participation. Participants in the optimisation group may benefit from improved preparation for surgery. The study also contributes to improving care for future patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status classification ≥ 3
* Age between 18 and 99 years
* All sexes
* Elective total hip or knee replacement with a waiting period of ≥ 8 weeks between surgical indication and surgery
* Ability to understand the nature, content, and procedures of the study and to provide written informed consent
* Written informed consent obtained prior to any study-related procedure

Exclusion Criteria:

* Pregnancy or active breastfeeding
* Severe trauma or major blood loss within 14 days prior to enrollment
* Participation in another pharmacological or interventional clinical study
* Contraindications to physical training
* Pre-existing diagnosis of moderate to severe dementia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2034-02-05 (Estimated); Study Completion 2034-02-05 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | From enrollment to the postoperative discharge from the hospital (9 to 25 weeks).
  Length of hospital stay (intensive care unit, recovery room, observation unit, general ward; date of discharge readiness and actual discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Sinner, MD, MBA, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria